CLINICAL TRIAL: NCT03128424
Title: Long Segment Lesion Peripheral Artery Revascularization Feasibility Study
Brief Title: TORUS I Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endologix (Industry)
Collaborators: PQ Bypass, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STP 185
Record Dates: First submitted 2016-08-29; First posted 2017-04-25 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- PQ Bypass Stent Graft System (Experimental): The PQ Bypass™ Stent Graft System is intended for patients with atherosclerotic lesions of the SFA
  Interventions: Device: PQ Bypass Stent Graft System

INTERVENTIONS:
Device: PQ Bypass Stent Graft System — The PQ Bypass™ Stent Graft System is indicated to improve luminal diameter in the treatment of patients with symptomatic de novo or restenotic native lesions or occlusions of the superficial femoral artery (SFA) and/or proximal popliteal artery, with reference vessel diameters of 5.0 to 6.7 mm and lesion lengths up to 180 mm.

SUMMARY:
The primary objective of the feasibility study is to evaluate the safety and effectiveness of the PQ Bypass Stent Graft System in the treatment of atherosclerotic lesions of the native superficial femoral artery (SFA) or the superficial femoral and proximal popliteal arteries.

DETAILED DESCRIPTION:
The primary safety endpoint for this study is freedom from a major adverse event (MAE) at 30 days post-procedure. An MAE is defined as TLR, amputation of the treated limb or death.

The primary effectiveness endpoint is defined as stent patency as evidenced by a peak systolic velocity ratio (PSVR) < 2.5 from DUS obtained within the 12-month visit window with no clinically-driven re-intervention within the stented segment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and of age of legal consent.
2. Women of child bearing potential must have a negative pregnancy test within 7 days prior to the index procedure.
3. Subject has lifestyle limiting claudication or rest pain (Rutherford Becker scale 2-4) with a resting ABI < 0.9. Resting TBI is utilized only if unable to reliably assess ABI. TBI must be <0.7. These assessments are required for the target limb, but both limbs are preferred.
4. A superficial femoral artery lesion with >50% stenosis or occlusion which requires treatment.
5. Stenotic lesion(s) or occluded length within the same vessel (one long or multiple serial lesions) ≥ 120mm to < 200mm.
6. Reference vessel diameter (RVD) ≥ 5.0mm and ≤ 6.7 mm, angiographically/CTA/MRA defined.
7. Patent popliteal artery 3 cm proximal to tibial plateau
8. At least 1 patent tibial artery to the foot (<50% stenosis)
9. The target lesion(s) can be successfully crossed with a guide wire and dilated.
10. Poor aortoiliac or common femoral "inflow" (i.e. angiographically defined >50% stenosis of the iliac or common femoral artery) that would be deemed inadequate to support a successful treatment of the target lesion without prior treatment. Adequate aortoiliac or common femoral "inflow" is defined as <30% stenosis after either PTA or stenting of the inflow lesion. After treatment of the inflow lesion, the residual pressure gradient across the target lesion will be obtained and if the peak to peak pressure gradient is < 20mmHg, the subject will be included in the study.
11. A subject with bilateral obstructive SFA disease is eligible for enrollment into the study. The contra-lateral procedure should not be done until at least 30 days after the index procedure (staged); however, if contra-lateral treatment is performed prior to treatment of the target lesion, the waiting period will be at least 30 days prior to the index procedure.
12. The subject is eligible for standard surgical repair, if necessary.
13. A subject who requires a coronary intervention should have it performed at least 30 days prior or 30 days post the treatment of the target lesion.
14. Subject must provide written informed consent.
15. Subject must be willing to comply with the specified follow-up evaluation schedule.

Exclusion Criteria:

1. Age greater than 90
2. Thrombophlebitis or deep venous thrombus, within the previous 30 days.
3. Receiving dialysis or immunosuppressant therapy within the previous 30 days.
4. Thrombolysis of the target vessel within 72 hours prior to the index procedure, where complete resolution of the thrombus was not achieved.
5. Stroke within the previous 90 days.
6. Ipsilateral femoral aneurysm or aneurysm in the SFA or popliteal artery.
7. Required stent placement via a popliteal approach.
8. Procedures which are pre-determined to require stent-in-stent placement to obtain patency, such as in-stent restenosis.
9. Significant vessel tortuosity or other parameters prohibiting access to the lesion or 90° tortuosity which would prevent delivery of the stent device.
10. Required stent placement within 1 cm of a previously deployed stent.
11. Known allergies to any of the following: aspirin and clopidogrel bisulfate (Plavix®), ticlopidine (Ticlid ®),and prasugrel (Effient®); heparin; Nitinol (nickel titanium); or contrast agent, that cannot be medically managed.
12. Presence of thrombus prior to crossing the lesion.
13. Known or suspected active infection at the time of the procedure.
14. Use of cryoplasty, laser, or atherectomy devices in the target vessel at the time of index procedure.
15. Restenotic lesion that had previously been treated by atherectomy, laser or cryoplasty within 3 months of the index procedure.
16. History of neutropenia, coagulopathy, or thrombocytopenia that was unexplained or is considered to be at risk for reoccurrence.
17. Known bleeding or hypercoagulability disorder or significant anemia (Hb<8.0) that cannot be corrected.
18. Subject has the following laboratory values: a. platelet count less than 80,000/μL, b. international normalized ratio (INR) greater than 1.5, c. serum creatinine level greater than 2.0 mg/dL.
19. Subject requires general anesthesia for the procedure.
20. Major distal amputation (above the transmetatarsal) in the study or non-study limb.
21. Patient has had a revascularization procedure on the target limb within 30 days of the planned index procedure
22. Patient has a planned amputation of the target limb
23. Previous bypass surgery on the target limb
24. Subject is pregnant or plans to become pregnant during the study.
25. Subject has a co-morbid illness that may result in a life expectancy of less than 1 year.
26. Subject is participating in an investigational study of a new drug, biologic or device at the time of study screening other than a PQ Bypass study.

NOTE: Subjects who are participating in the long term follow-up phase of a previously investigational and now CE marked product are not excluded by this criterion.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2021-09 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PQ Bypass Stent Graft System
Started | 60
Completed | 55
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | PQ Bypass Stent Graft System
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 30
  Austria | 1
  Latvia | 20
  Poland | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Freedom From a Major Adverse Event (MAE)
Description: Freedom from a MAE as defined as target lesion revascularization (TLR), amputation of the treated limb or death.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | PQ Bypass Stent Graft System
Number analyzed (Participants) | 60
Participants | 60

2. Primary Outcome: Primary Effectiveness
Description: The primary effectiveness endpoint is defined as stent patency as evidenced by a peak systolic velocity ratio (PSVR) < 2.5 from DUS obtained within the 12- month visit window with no clinically driven re-intervention within the stented segment
Time Frame: 12 Month
Population: Through 12 months, 50 subjects provided data on both PSVR and clinically driven re-intervention. Subjects with Absolute peak systolic velocity (PSV) numbers and no PSVR ratio were included in the primary patency assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | PQ Bypass Stent Graft System
Number analyzed (Participants) | 50
Participants | 38

3. Secondary Outcome: Technical Success
Description: Acute technical successdefined as : successful delivery, access and placement of the investigation devies and successful removal of the delivery system
Time Frame: Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | PQ Bypass Stent Graft System
Number analyzed (Participants) | 60
Participants | 60

4. Secondary Outcome: Lesion Success
Description: Clinically Driven Target Lesion Revascularization (CD-TLR)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | PQ Bypass Stent Graft System
Number analyzed (Participants) | 60
Participants
  12 months Rate of CD-TLR | 4
  12 Month Freedom from CD-TLR | 56

5. Secondary Outcome: Major Adverse Event (MAE) 6 Month
Description: A Major Adverse Event (MAE) is defined as all cause mortality, target limb major amputation, and clinically driven target lesion revascularization (CD-TLR).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | PQ Bypass Stent Graft System
Number analyzed (Participants) | 60
Participants | 1

6. Secondary Outcome: Major Adverse Event (MAE) 12 Months
Description: An MAE is defined as target lesion revascularization (TLR), amputation of the treated limb or death.
Time Frame: 12 month
Measure: Count of Participants; unit: Participants
Arm/Group | PQ Bypass Stent Graft System
Number analyzed (Participants) | 60
Participants | 5

7. Secondary Outcome: TORUS Stent Fracture, Migration, and Separation
Description: Stent Fracture, Migration, and Separation
Time Frame: 12 Month
Measure: Count of Participants; unit: Participants
Arm/Group | PQ Bypass Stent Graft System
Number analyzed (Participants) | 60
Participants | 0

ADVERSE EVENTS:
Time Frame: 24 Months
Description: Adverse events were reviewed by an independent Medical Monitor. MedDRA Lower-Level Terms (LLTs) were assigned by a certified MedDRA coder. The LLTs were mapped to their corresponding Preferred Terms (PTs) and System Organ Categories (SOCs).
Arm/Group | PQ Bypass Stent Graft System
All-Cause Mortality (participants affected / at risk) | 2/60
Serious Adverse Events (participants affected / at risk) | 31/60
Other Adverse Events (participants affected / at risk) | 30/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PQ Bypass Stent Graft System (N=60)
Cardiac disorders (Cardiac disorders) | 6
Eye disorders (Eye disorders) | 1
Gastrointestinal disorders (Gastrointestinal disorders) | 4
General disorders and administration site conditions (General disorders) | 24
Immune system disorders (Immune system disorders) | 1
Infections and infestations (Infections and infestations) | 2
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant, and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nervous system disorders (Nervous system disorders) | 2
Respiratory, thoracic, and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2
Surgical and medical procedures (Surgical and medical procedures) | 3
Vascular disorders (Vascular disorders) | 10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PQ Bypass Stent Graft System (N=60)
Cardiac disorders (Cardiac disorders) | 5
General disorders and administration site conditions (General disorders) | 21
Infections and infestations (Infections and infestations) | 3
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 3
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 3
Nervous system disorders (Nervous system disorders) | 1
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1
Surgical and medical procedures (Surgical and medical procedures) | 1
Vascular disorders (Vascular disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT03128424/Prot_SAP_000.pdf